CLINICAL TRIAL: NCT00140868
Title: Outcome of Palliative Management of Malignant Large Bowel Obstruction With Colorectal Stents or Surgery
Brief Title: Outcome of Palliative Management of Malignant Large Bowel Obstruction w/Colorectal Stents or Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 02-125
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Large Bowel Obstruction
Keywords: Colonic Pseudo-Obstruction; Large bowel obstruction; Stents; Laparotomy; Palliative Surgery; Surgery, Palliative; Palliative Therapy
MeSH Terms: conditions — Colonic Pseudo-Obstruction

INTERVENTIONS:
Device: Luminal stents
Procedure: Minimally Invasive Surgical Bowel Diversion

SUMMARY:
The purpose of this study is to assess quality of life and bowel symptoms after treatment.The main objective is to compare the effect on quality of life of minimally invasive bowel surgery and endoscopic stent placement in the treatment of malignant large bowel obstruction.

DETAILED DESCRIPTION:
Large bowel obstruction is a common presentation among cancer patients, including those with non-colorectal malignancies. This study will evaluate patients with malignant large bowel obstruction who undergo palliative treatment with minimally invasive surgical diversion or endoscopic colorectal stent placement, in terms quality of life, symptom relief from bowel obstruction, and treatment-related complications. Assessments in changes in quality of life and symptom relief over time for each group will be done.

Traditionally malignant bowel obstruction is treated with surgery. In the last decade, creation of an ostomy can be completed with minimally invasive surgery, which reduces morbidity, mortality, and recovery time.wishes.

In the last several years, endoscopically inserted colorectal stents have emerged as an option for palliative treatment. This involves a simple procedure, often completed on an outpatient basis. This allows the intestinal lumen to remain open without the need for surgery.

* Primary Objective: is to compare the effect on quality of life of minimally invasive surgical bowel diversion and endoscopic stent placement in the treatment of malignant large bowel obstruction.
* Secondary Objectives: are to evaluate the symptom response (including abdominal pain, distention, bowel frequency and consistency, and nausea and emesis) and complication rate of treatment of malignant large bowel obstruction with endoscopic stent placement or minimally invasive surgical bowel diversion.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18 years of age
* presentation of large bowel obstruction based on clinical symptoms AND an imaging study.
* clinical symptoms: one of : progressive constipation, multiple small liquid bowel movements daily, abdominal distention, abdominal pain or nausea and vomiting.
* imaging study: one of: CT scan, barium or gastrograffin enema, flexible sigmoidoscopy or colonoscopy, showing any degree of colonic narrowing by tumor.
* large bowel obstruction due to stage IV colorectal cancer unresectable for cure OR unresectable local-regional colorectal cancer OR unresectable extra-colonic cancer (such as gastric, ovarian, prostate, pancreatic cancers).
* ability to give informed consent, indicating the investigational nature of this study in keeping with the policies of Memorial Sloan-Kettering Cancer Center.

Exclusion Criteria:

* presence of acute bowel perforation
* presence of a second synchronous large or small bowel obstruction site
* contra-indication to stent placement:
* obstruction greater than 12 cm in length (ie precluding treatment with one stent)
* obstruction located within 2 cm of dentate line
* contra-indication to laparoscopy:
* presence of MI, unstable angina, or CVA in the previous four weeks
* tense ascites
* uncorrectable coagulopathy
* prior abdominal surgery with known prohibitive adhesions
* prior PALLIATIVE treatment of malignant large bowel obstruction with surgery or stent
* inability to speak or read English, or other impairment which causes an inability to complete the quality of life questionnaires
* unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2002-12; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Primary objective: compare the effect on quality of life of minimally invasive surgical bowel diversion and endoscopic stent placement in the treatment of malignant large bowel obstruction.

SECONDARY OUTCOMES:
Secondary objectives:the symptom response and complication rate of treatment of malignant large bowel obstruction with endoscopic stent placement or minimally invasive surgical bowel diversion

CONTACTS AND LOCATIONS:
Overall Officials: Hans Gerdes, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org